CLINICAL TRIAL: NCT01098955
Title: Smoking Cessation Treatment for Head & Neck Cancer Patients: Acceptance and Commitment Therapy
Brief Title: Smoking Cessation Treatment for Head & Neck Cancer Patients
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0362; NCI-2011-02004 (Registry Identifier: NCI CTRP); 1R01CA120153-01A2 (NIH)
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer; Smoking Cessation
Keywords: Cancer; Smoking Cessation Treatment; Acceptance and Commitment Therapy; ACT Theory; Motivational and Behavioral Counseling; MBC; abstinence; Varenicline; Chantix
MeSH Terms: conditions — Head and Neck Neoplasms; Smoking Cessation; Neoplasms | interventions — Acceptance and Commitment Therapy; Behavior Therapy; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACT Group 1 (Experimental): Acceptance and Commitment Therapy (ACT). Varenicline 2 mg daily for 12 weeks.
  Interventions: Behavioral: Acceptance and Commitment Therapy; Drug: Varenicline
- MBC Group 2 (Experimental): Motivational and Behavioral Counseling (MBC). Varenicline 2 mg daily for 12 weeks.
  Interventions: Behavioral: Motivational and Behavioral Counseling; Drug: Varenicline

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — 6 x 60-minute counseling sessions delivered over a 5-week period
  Arms: ACT Group 1
Behavioral: Motivational and Behavioral Counseling — 6 x 60-minute counseling sessions delivered over a 5-week period
  Arms: MBC Group 2
Drug: Varenicline — 2 mg daily for 12 weeks
  Other Names: Chantix

SUMMARY:
This is Part 1 of a 2-part research study. The goal of this part of the study is to plan and test an investigational type of counseling called Acceptance and Commitment Therapy, for use in patients who have or had head and neck cancer, lung cancer, breast cancer, gastrointestinal cancer, or genitourinary cancer.

This part of the study is also designed to train the study counselors how to perform Acceptance and Commitment Therapy.

In this part of the study, participants will either receive Acceptance and Commitment Therapy or the standard type of counseling, called Motivational and Behavioral Counseling.

This is Part 2 of a 2-part research study. In both parts of the study, participants receive either an investigational type of counseling (Acceptance and Commitment Therapy) or a standard type of counseling (Motivational and Behavioral Counseling). Part 1 was also designed to train the study counselors how to perform Acceptance and Commitment Therapy.

The goal of Part 2 is to compare Acceptance and Commitment Therapy against Motivational and Behavioral Counseling. Researchers want to learn which type of counseling may be more effective in helping patients to stop smoking. These types of counseling will be tested in patients who have or had head and neck cancer, lung cancer, breast cancer, gastrointestinal cancer, or genitourinary cancer.

DETAILED DESCRIPTION:
Part 1:

Counseling to Quit Smoking Acceptance and Commitment Therapy is designed to help patients change the way they respond to feelings and thoughts that cause them to want to smoke. It is also designed to help increase patients' ability to tolerate negative feelings about cancer, and to increase patients' commitment to other goals that are related to what they value in life.

Motivational and Behavioral Counseling is designed to help patients increase their motivation to quit smoking. It is also designed to help patients develop skills and behaviors that will help them cope with situations when they want to smoke.

Baseline Tests:

If you are found to be eligible to take part in the pilot study, you will have additional "baseline" tests. This will include a series of questionnaires, which will take about 30 minutes to complete, and a saliva test. These tests will be done at the same visit as the screening tests.

You will fill out 10 or 11 questionnaires that relate to:

* smoking
* any symptoms of nicotine dependence and withdrawal
* your feelings and thoughts in response to urges to smoke
* your confidence in your ability to quit smoking
* your reasons for quitting smoking
* your mood
* your use of alcohol
* the general quality of your life
* any effects of cancer on your ability to take part in everyday activities
* your response to stressful events in your life

Saliva will be collected to check for a chemical called cotinine. This test will help researchers measure how much you are smoking. To collect saliva, a cotton swab will be placed in your mouth for several minutes.

The information you provide in the Tobacco Treatment Program (TTP) questionnaires regarding anxiety, depression, alcohol use, sleeping difficulties, smoking withdrawal symptoms, nicotine dependence and smoking will be used for this study, so that you do not have to fill out these questionnaires twice. Physical data that you provided to the TTP (such as breath samples, blood pressure, heart rate and weight) will also be used in this study, so that it does not have to be collected twice.

Study Groups:

You will be assigned to 1 of 2 groups. The group you are in will be decided based on the study counselors' training schedules and other study needs.

* Group 1 will receive Acceptance and Commitment Therapy.
* Group 2 will receive Motivational and Behavioral Counseling.

You will receive a booklet that describes the type of counseling you will receive.

Varenicline as Standard Care:

Participants in both groups will receive varenicline through the Tobacco Treatment Program. Varenicline is designed to imitate the effects that nicotine has on the body. This may reduce cigarette cravings and help people quit smoking.

As part of your counseling sessions, you will be counseled to help you make a plan to quit smoking and to set a quit date. The quit date may be scheduled for about 3 weeks after your screening/baseline visit.

You will be provided with a 10-week supply of varenicline. Your first dose will be at least 2 weeks before the quit date, and you will continue taking varenicline until 8 weeks after the quit date. You will take it by mouth, 2 times a day.

Varenicline is the standard drug that is given in the Tobacco Treatment Program.

The Tobacco Treatment Program staff will discuss the risks of varenicline with you.

Counseling Visits:

You will have 6 visits with a study counselor during the 12 weeks after your screening/baseline visit.

At every visit:

* You will receive counseling that will last about an hour.
* You will fill out 5-8 questionnaires about smoking, mood, alcohol use, quality of life, and coping. This should take about 20-30 minutes.
* You will be asked about any changes in the drugs or other treatments you may be receiving.
* You will be asked about how you took varenicline.
* You will be given homework assignments that will help you practice the skills that you learn during the visits. There will be 1 or 2 homework assignments per week, and each assignment will take about 30 minutes.

At your last counseling visit (Counseling Visit 6), you will be asked questions about how satisfied you may be with the study counseling. Also at this visit, the research staff may ask you to provide a saliva sample that will be used to measure if and how much you have smoked.

If you do not complete all 6 of the counseling sessions, the research staff will call and ask you what made it difficult for you to complete the counseling sessions.

Videotaping:

Each of the counseling visits will be videotaped. The videotapes will be used to help the research staff make sure that the study counselors are following the correct therapy procedures.

The videotapes will probably be saved for 2 years and then destroyed. However, it is possible that these videotapes will be saved for a longer period of time.

Only the research staff, study counselors, and study consultants will be allowed to watch the tapes. The study consultants will review the tapes and rate how well the study counselors follow therapy procedures. One consultant is an associate professor at the University of Mississippi. The other consultant is a research scientist at the University of Texas. Another consultant is an assistant professor at University of Washington. All are collaborators for this study and part of the research team.

Safety Procedures:

Quitting smoking may cause side effects affecting your mental and emotional health. For your safety, the study counselor and study chair will be looking for any signs that you may be having these side effects.

If the study counselor or study chair think that you may be having emotional difficulties or depression, they may decide to recommend that you be treated for it.

If they believe you are at risk of being a danger to yourself, you will be contacted by the study chair right away and if appropriate, you will be referred to meet with the Tobacco Treatment Program psychiatrist (mental health doctor).

Follow-Up Visit:

You will have a follow-up visit at 3 months after your quit date. You will complete most of the same questionnaires that you completed at the screening/baseline visit, and this should take about 30 minutes. The research staff also may ask you to provide a saliva sample that will be used to measure if and how much you have smoked.

Length of Study:

Your participation in this study will be over after your follow-up visit.

This is an investigational study. Acceptance and Commitment Therapy is investigational, and Motivational and Behavioral Counseling is standard.

Varenicline is FDA approved and commercially available to help people stop smoking.

Up to 108 patients will take part in this study. This includes 12 participants who are interviewed before Part 1 opens, 20 participants in Part 1, and 76 participants in Part 2. All will be enrolled at MD Anderson.

Part 2:

Acceptance and Commitment Therapy is designed to help patients change the way they respond to feelings and thoughts that cause them to want to smoke. It is also designed to help increase patients' ability to tolerate negative feelings about cancer, and to increase patients' commitment to other goals that are related to what they value in life.

Motivational and Behavioral Counseling is designed to help patients increase their motivation to quit smoking. It is also designed to help patients develop skills and behaviors that will help them cope with situations when they want to smoke.

Baseline Tests:

If you are found to be eligible to take part in this study, you will have additional "baseline" tests. This will include a series of questionnaires, which will take about 30 minutes to complete, and a saliva test. These tests will be done at the same visit as the screening tests.

You will fill out 10 or 11 questionnaires that relate to:

* smoking
* any symptoms of nicotine dependence and withdrawal
* your feelings and thoughts in response to urges to smoke
* your confidence in your ability to quit smoking
* your reasons for quitting smoking
* your mood
* your use of alcohol
* the general quality of your life
* any effects of cancer on your ability to take part in everyday activities
* your response to stressful events in your life

Saliva will be collected to check for a chemical called cotinine. This test will help researchers measure how much you are smoking. To collect saliva, a cotton swab will be placed in your mouth for several minutes.

The information you provide in the Tobacco Treatment Program (TTP) questionnaires regarding anxiety, depression, alcohol use, sleeping difficulties, smoking withdrawal symptoms, nicotine dependence and smoking will be used for this study, so that you do not have to fill out these questionnaires twice. Physical data that you provided to the TTP (such as breath samples, blood pressure, heart rate and weight) will also be used in this study, so that it does not have to be collected twice. Some of the data you provide to this study regarding mood, nicotine withdrawal, and smoking will be provided to the TTP so that it does not have to be collected twice.

Study Groups:

You will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. There is an equal chance that you will be assigned to either group.

* Group 1 will receive Acceptance and Commitment Therapy.
* Group 2 will receive Motivational and Behavioral Counseling.

You will receive a booklet that describes the type of counseling you will receive.

Varenicline as Standard Care:

Participants in both groups will receive varenicline through the Tobacco Treatment Program.

As part of your counseling sessions, you will be counseled to help you make a plan to quit smoking and to set a quit date, if you so choose.

You will be provided with 10 weeks of medication. You will take it by mouth, up to 2 times a day.

Varenicline is the standard drug that is given in the Tobacco Treatment Program. The Tobacco Treatment Program staff will discuss the risks of varenicline with you.

Counseling Visits:

You will have 6 visits with a study counselor during the 12 weeks after your screening/baseline visit.

At every visit:

* You will receive counseling that will last about an hour.
* You will fill out 5-8 questionnaires about smoking, mood, alcohol use, quality of life, and coping. This should take about 20-30 minutes.
* You will be asked about any changes in the drugs or other treatments you may be receiving.
* You will be asked about how you took varenicline.
* You will be given homework assignments that will help you practice the skills that you learn during the visits. There will be 1 or 2 homework assignments per week, and each assignment will take about 30 minutes.

At your last counseling visit (Counseling Visit 6), the research staff may ask you to provide a saliva sample that will be used to measure if and how much you have smoked.

Videotaping:

Each of the counseling visits will be videotaped. The videotapes will be used to help the research staff make sure that the study counselors are following the correct therapy procedures.

The videotapes will probably be saved for 2 years and then destroyed. However, it is possible that these videotapes will be saved for a longer period of time.

Only the research staff, study counselors, and study consultants will be allowed to watch the tapes. The study consultants will review the tapes and rate how well the study counselors follow therapy procedures. One consultant is an associate professor at the University of Mississippi, one consultant is a research scientist at the University of Texas, and the last consultant is an assistant professor at University of Washington. All are collaborators for this study and part of the research team.

Safety Procedures:

Quitting smoking may cause side effects affecting your mental and emotional health. For your safety, the study counselor and study chair will be looking for any signs that you may be having these side effects.

If the study counselor or study chair think that you may be having emotional difficulties or depression, they may decide to recommend that you be treated for it.

If they believe you are at risk of being a danger to yourself, you will be contacted by the study chair right away and if appropriate, you will be referred to meet with the Tobacco Treatment Program psychiatrist (mental health doctor).

Follow-Up Visits:

You will have follow-up visits at 3 and 6 months after your quit date. You will complete most of the same questionnaires that you completed at the screening/baseline visit, and this should take about 30 minutes. At these visits, the research staff may ask you to provide a saliva sample that will be used to measure if and how much you have smoked.

Length of Study:

Your participation in this study will be over after your second follow-up visit.

This is an investigational study. Acceptance and Commitment Therapy is investigational, and Motivational and Behavioral Counseling is standard.

Varenicline is FDA approved and commercially available to help people stop smoking.

Up to 108 patients will take part in this study. This includes 12 participants who are interviewed before Part 1 opens, 20 participants in Part 1, and 76 participants in Part 2. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Current or history of head and neck, lung, breast, gastrointestinal, or genitourinary cancer
2. Age 18 or older
3. Smoking 1 cigarette or more per day at screening visit
4. English speaking and have a telephone
5. Willing to provide informed consent and agree to all assessments and study procedures
6. Recommended for and agreed to treatment with varenicline through the Tobacco Treatment Program
7. Plan to receive treatment for head and neck, lung, breast, gastrointestinal, or genitourinary cancer, currently undergoing treatment, or in follow-up care at M.D. Anderson Cancer Center

Exclusion Criteria:

1. Anticipated hospitalization of 2 weeks or longer
2. Planned total laryngectomy
3. Current use of bupropion, nortriptyline, clonidine or nicotine replacement therapy
4. Currently receiving other forms of smoking cessation treatment
5. Severe levels of depressive symptoms, vegetative symptoms, and/or symptoms related to psychiatric disorders that place participant at risk for harm or require immediate treatment
6. Currently pregnant or lactating
7. Has received treatment in the TTP
8. History or/current medical condition, or any other factor that , in the judgment of the PI would likely preclude completion of study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-03-24 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence Rate | Baseline up to 6 weeks
  Participants will be assessed on a variety of interview, self-report, and biochemical measures at baseline, at key points during treatment (including end of treatment), and at 14-, and 26-weeks after the targeted quit date

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blalock, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org